CLINICAL TRIAL: NCT06113887
Title: The Effect of Acceptance and Commitment Therapy Based Psychoeducation on Psychological Flexibility and Impulsivity Levels in Bipolar Disorder Patients
Brief Title: The Effect of Acceptance and Commitment of Bipolar Disorder Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Kubra TOHUMCU, Principal Investigator, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Gaziantep University KTOHUMCU
Record Dates: First submitted 2023-09-21; First posted 2023-11-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Psychological Flexibility; Impulsivity; Acceptance and Commitment Therapy; Psychoeducation
MeSH Terms: conditions — Bipolar Disorder; Impulsive Behavior

STUDY DESIGN:
Intervention Model Description: A total of 10 groups, 5 intervention groups and 5 control groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- intervention group 1 in which psychoeducation based on acceptance and commitment therapy was applied (Experimental): Personal Information Form, Psychological Flexibility Scale and Barratt Impulsivity Scale -11 Short Form (BIS-11-SF) pre-tests will be applied. After the pre-test, acceptance and stability-based psychoeducation consisting of 8 modules will be implemented once a week as a single module. Each session of the acceptance and stability therapy-based psychoeducation, which will last 8 weeks in total, will be implemented for 45-60 minutes. Immediately after the training sessions are completed, the post-test; Psychological Flexibility Scale and Barratt Impulsivity Scale -11 Short Form (BIS-11-SF) will be administered. A follow-up test will be administered one month after the post-test, i.e. in the 12th week.
  Interventions: Other: psychoeducation based on acceptance and commitment therapy
- Control group 1 (No Intervention): Personal Information Form, Psychological Flexibility Scale and Barratt Impulsivity Scale -11 Short Form (BIS-11-SF) pre-tests will be applied. After the pre-test is administered, post-test will be administered in the 8th week and follow-up tests will be administered in the 12th week without any intervention.
- Intervention group 2 in which psychoeducation based on acceptance and commitment therapy was applied (Experimental): Personal Information Form, Psychological Flexibility Scale and Barratt Impulsivity Scale -11 Short Form (BIS-11-SF) pre-tests will be applied. After the pre-test, acceptance and stability-based psychoeducation consisting of 8 modules will be implemented once a week as a single module. Each session of the acceptance and stability therapy-based psychoeducation, which will last 8 weeks in total, will be implemented for 45-60 minutes. Immediately after the training sessions are completed, the post-test; Psychological Flexibility Scale and Barratt Impulsivity Scale -11 Short Form (BIS-11-SF) will be administered. A follow-up test will be administered one month after the post-test, i.e. in the 12th week.
  Interventions: Other: psychoeducation based on acceptance and commitment therapy
- Control group 2 (No Intervention): Personal Information Form, Psychological Flexibility Scale and Barratt Impulsivity Scale -11 Short Form (BIS-11-SF) pre-tests will be applied. After the pre-test is administered, post-test will be administered in the 8th week and follow-up tests will be administered in the 12th week without any intervention.
- Intervention group 3 in which psychoeducation based on acceptance and commitment therapy was applied (Experimental): Personal Information Form, Psychological Flexibility Scale and Barratt Impulsivity Scale -11 Short Form (BIS-11-SF) pre-tests will be applied. After the pre-test, acceptance and stability-based psychoeducation consisting of 8 modules will be implemented once a week as a single module. Each session of the acceptance and stability therapy-based psychoeducation, which will last 8 weeks in total, will be implemented for 45-60 minutes. Immediately after the training sessions are completed, the post-test; Psychological Flexibility Scale and Barratt Impulsivity Scale -11 Short Form (BIS-11-SF) will be administered. A follow-up test will be administered one month after the post-test, i.e. in the 12th week.
  Interventions: Other: psychoeducation based on acceptance and commitment therapy
- Control group 3 (No Intervention): Personal Information Form, Psychological Flexibility Scale and Barratt Impulsivity Scale -11 Short Form (BIS-11-SF) pre-tests will be applied. After the pre-test is administered, post-test will be administered in the 8th week and follow-up tests will be administered in the 12th week without any intervention.
- Intervention group 4 in which psychoeducation based on acceptance and commitment therapy was applied (Experimental): Personal Information Form, Psychological Flexibility Scale and Barratt Impulsivity Scale -11 Short Form (BIS-11-SF) pre-tests will be applied. After the pre-test, acceptance and stability-based psychoeducation consisting of 8 modules will be implemented once a week as a single module. Each session of the acceptance and stability therapy-based psychoeducation, which will last 8 weeks in total, will be implemented for 45-60 minutes. Immediately after the training sessions are completed, the post-test; Psychological Flexibility Scale and Barratt Impulsivity Scale -11 Short Form (BIS-11-SF) will be administered. A follow-up test will be administered one month after the post-test, i.e. in the 12th week.
  Interventions: Other: psychoeducation based on acceptance and commitment therapy
- Control group 4 (No Intervention): Personal Information Form, Psychological Flexibility Scale and Barratt Impulsivity Scale -11 Short Form (BIS-11-SF) pre-tests will be applied. After the pre-test is administered, post-test will be administered in the 8th week and follow-up tests will be administered in the 12th week without any intervention.
- Intervention group 5 in which psychoeducation based on acceptance and commitment therapy was applied (Experimental): Personal Information Form, Psychological Flexibility Scale and Barratt Impulsivity Scale -11 Short Form (BIS-11-SF) pre-tests will be applied. After the pre-test, acceptance and stability-based psychoeducation consisting of 8 modules will be implemented once a week as a single module. Each session of the acceptance and stability therapy-based psychoeducation, which will last 8 weeks in total, will be implemented for 45-60 minutes. Immediately after the training sessions are completed, the post-test; Psychological Flexibility Scale and Barratt Impulsivity Scale -11 Short Form (BIS-11-SF) will be administered. A follow-up test will be administered one month after the post-test, i.e. in the 12th week.
  Interventions: Other: psychoeducation based on acceptance and commitment therapy
- Control group 5 (No Intervention): Personal Information Form, Psychological Flexibility Scale and Barratt Impulsivity Scale -11 Short Form (BIS-11-SF) pre-tests will be applied. After the pre-test is administered, post-test will be administered in the 8th week and follow-up tests will be administered in the 12th week without any intervention.
- Intervention group 6 in which psychoeducation based on acceptance and commitment therapy was applied (Experimental): Personal Information Form, Psychological Flexibility Scale and Barratt Impulsivity Scale -11 Short Form (BIS-11-SF) pre-tests will be applied. After the pre-test, acceptance and stability-based psychoeducation consisting of 8 modules will be implemented once a week as a single module. Each session of the acceptance and stability therapy-based psychoeducation, which will last 8 weeks in total, will be implemented for 45-60 minutes. Immediately after the training sessions are completed, the post-test; Psychological Flexibility Scale and Barratt Impulsivity Scale -11 Short Form (BIS-11-SF) will be administered. A follow-up test will be administered one month after the post-test, i.e. in the 12th week.
  Interventions: Other: psychoeducation based on acceptance and commitment therapy
- Control group 6 (No Intervention): Personal Information Form, Psychological Flexibility Scale and Barratt Impulsivity Scale -11 Short Form (BIS-11-SF) pre-tests will be applied. After the pre-test is administered, post-test will be administered in the 8th week and follow-up tests will be administered in the 12th week without any intervention.

INTERVENTIONS:
Other: psychoeducation based on acceptance and commitment therapy — Acceptance and Commitment Therapy Based Psychoeducation will be applied to the patients in the intervention group in the form of group education (consisting of 5-7 people), one session per week for eight weeks; no intervention will be applied to the control group.
  Arms: Intervention group 2 in which psychoeducation based on acceptance and commitment therapy was applied; Intervention group 3 in which psychoeducation based on acceptance and commitment therapy was applied; Intervention group 4 in which psychoeducation based on acceptance and commitment therapy was applied; Intervention group 5 in which psychoeducation based on acceptance and commitment therapy was applied; Intervention group 6 in which psychoeducation based on acceptance and commitment therapy was applied; intervention group 1 in which psychoeducation based on acceptance and commitment therapy was applied

SUMMARY:
This study will be conducted to determine the effect of acceptance and commitment therapy-based psychoeducation on psychological flexibility and impulsivity levels in patients with bipolar disorder. This study was planned as a randomised controlled experimental study. The study will be conducted with 60 patients (Intervention: 30, Control: 30) in the euthymic stage diagnosed with bipolar disorder who applied to Adıyaman Besni State Hospital psychiatry outpatient clinic using randomisation method. "Introductory Information Form" about socio-demographic characteristics, "Psychological Flexibility Scale" and "Barratt Impulsivity Scale -11 Short Form" will be used for data collection. Acceptance and Commitment Therapy Based Psychoeducation will be applied to the patients in the intervention group in the form of group education (consisting of 5-7 people), one session per week for eight weeks; no intervention will be applied to the control group. Pre-tests will be applied to the patients in the intervention and control groups just before the training, post-test will be applied to the intervention group immediately after the training sessions are completed, and follow-up test will be applied one month after the post-test, i.e. in the 12th week. After the pre-test was applied to the control group, the post-test will be applied in the 8th week and the follow-up test will be applied in the 12th week without any intervention. Repeated Measures Analysis of Variance was used to compare the scale scores and Fisher Least Significant Difference test was used for multiple comparisons of Group*Time interaction. Permission was obtained from the University Ethics Committee, the relevant institution and the individuals participating in the study.

DETAILED DESCRIPTION:
INTRODUCTION Bipolar disorder ranks sixth among the causes of disability in the world due to its serious individual, family, social and economic burden. In patients with bipolar disorder, functioning may be impaired even in the euthymic period and psychopathological dimensions such as impulsivity negatively affect functioning. Impulsivity is defined as taking action quickly without thinking beforehand or making a conscious decision, in other words, exhibiting behaviour without sufficient thought. Impulsivity has a central role in the etiopathogenesis of mood disorders. One of the reasons for the low functionality and quality of life of individuals diagnosed with bipolar disorder is that these individuals have lower psychological flexibility than healthy individuals. The concept of psychological flexibility is the ability of an individual to consciously connect with the present moment and to act in line with his/her values. Psychological flexibility is the cornerstone of healthy personal and social functioning. However, many forms of psychopathology lack these resilience processes. Interventions to increase resilience help both sick and healthy individuals and are believed to be an important force in increasing their effectiveness and satisfaction in life. Individuals with bipolar disorder are often disorganised in their daily lives, even when euthymic, and may also benefit from psychosocial treatments aimed at improving cognitive functioning to increase their ability to function in daily life.

Cognitive Behavioural Therapy is one of the important psychosocial interventions applied in bipolar disorder. The therapy model called Acceptance and Commitment Therapy is one of the leading therapy types among the third generation cognitive behavioural therapy approaches. The main aim of Acceptance and Commitment Therapy is to increase the general psychological flexibility of individuals. Psychological flexibility plays an important role in the etiology, course and clinical presentation of bipolar disorder, as in many psychiatric disorders. Treatment of impulsivity in patients with bipolar disorder is provided by pharmacotherapy and various psychotherapeutic approaches. People with high levels of psychological rigidity exhibit impulsive behaviours such as avoidance, escape or self-harm by turning to the use of psychoactive substances to reduce the intensity of their internal experiences that they define as negative or to get rid of them. Studies have shown the significant potential impact of Acceptance and Commitment Therapy in many mental health conditions, including mood disorders and psychotic symptoms. It is thought that the application of a psychoeducation programme based on acceptance and commitment therapy to individuals diagnosed with bipolar disorder may help to increase the psychological flexibility of these individuals and decrease impulsivity as a result of increased psychological flexibility. All developments related to the understanding of the etiology and treatment of impulsivity will make a significant contribution to the understanding of mental illnesses. As far as we can reach, there is no randomised controlled study in the literature in which the results of acceptance and commitment therapy-based psychoeducation interventions in individuals diagnosed with bipolar disorder have been published.

METHOD This research is a randomised controlled experimental study. The research is planned to be conducted in Adıyaman Besni State Hospital between November 2022 and November 2023. The population of the study will consist of individuals who applied to the Psychiatry Outpatient Clinic of Adıyaman Besni State Hospital on the dates of the study, who received outpatient treatment with the diagnosis of bipolar according to Diagnostic and Statistical Manual of Mental Disorders-5 and who were in the euthymic period according to the doctor's control. Using the randomisation method, 60 individuals diagnosed with bipolar disorder who meet the inclusion criteria, volunteer to participate in the study and apply on the data collection dates of the study will constitute the sample of the study. The research will be completed with a total of 60 patients (30 experimental, 30 control) by taking 30 individuals diagnosed with bipolar disorder into the experimental group and 30 individuals into the control group.

G Power programme was used to calculate the sample size. The data will be collected by the researcher Kübra Tohumcu by face-to-face interview technique in the training room of Adıyaman Besni State Hospital. The patients constituting the sample of the study will be directed to the researcher by the outpatient clinic doctor. The patients who will be directed to the researcher by the doctor will first be informed about the research and the patients who meet the inclusion criteria will be determined as experimental and control groups by randomisation method.

It is planned to apply Acceptance and Commitment Therapy Based Psychoeducation Programme to the patients to be included in the experimental group. Personal Information Form, Psychological Flexibility Scale and Barratt Impulsivity Scale -11 Short Form pre-tests will be applied to the patients in the experimental and control groups just before the training. In the first interview with the patients in the experimental group, information about the training will be given and training days and hours will be determined. Then, acceptance and stability-based psychoeducation consisting of 8 modules will be applied to the individuals in the experimental group once a week as a single module. Each session of acceptance and stability therapy-based psychoeducation, which will last for 8 weeks in total, will be 45-60 minutes. Sessions will consist of 5-7 people on average and will be held as group training. The groups will be closed groups and new patients will not be included in the groups after the training sessions begin. In order to complete the sufficient number of data, new groups will be formed with the patients recruited later. Immediately after the training sessions are completed, the post-test; Psychological Flexibility Scale and Barratt Impulsivity Scale -11 Short Form will be applied to the experimental group. One month after the post-test, i.e. in the 12th week, a follow-up test will be applied to the experimental group. The control group will be administered the post-test at the 8th week and the follow-up test at the 12th week without any intervention after the pre-test.

Data Collection Tools Personal Information Form: This form, organised by the researchers, includes 17 questions to determine the demographic information of the participants.

Psychological Flexibility Scale: The scale is a 7-point Likert-type scale (1=strongly disagree, 7=strongly agree) consisting of 28 items. The scale has 5 sub-dimensions: "Values and behaviour in line with values", "Being in the moment", "Acceptance", "Contextual Self" and "Dissociation". When evaluating the scale, 6 different sub-scores can be obtained, including the scores obtained from each sub-dimension and the total score. The lowest score to be obtained from the scale is 28 and the highest score is 196. High scores obtained from the scale indicate the high psychological flexibility of individuals.

Barratt Impulsivity Scale -11 Short Form: The scale consists of a total of 15 items and three subscales. These subscales are lack of planning, motor impulsivity and attention impulsivity. The items in the scale are evaluated using a 4-point Likert-type scale (1=rarely/never, 4=almost always/always).

Data Analysis: The data obtained from the study will be analysed in Statistical Package for Social Sciences 22 package programme. Repeated Measures Analysis of Variance was used to compare the scale scores and Fisher Least Significant Difference test was used for multiple comparisons of Group*Time interaction.

ELIGIBILITY:
Inclusion Criteria:

* • To be receiving outpatient treatment with the diagnosis of Bipolar Disorder according to DSM-5

  * Being in euthymic mood according to the doctor's control at the time of the interview
  * Having no problem in understanding and speaking Turkish
  * Being literate
  * Being in the 18-65 age group
  * Not having undergone such training for the last 1 year

Exclusion Criteria:

* • Presence of serious sensory and cognitive disabilities that would prevent answering the questionnaire

  * Refusal to participate in the study after being informed
  * Having another psychiatric diagnosis in addition to the diagnosis of bipolar disorder
  * Having an attack period during the education process

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
The effect of psychoeducation based on acceptance and commitment therapy on psychological flexibility level in bipolar disorder patients | up to 12 weeks
  The effect of psychoeducation based on acceptance and commitment therapy on psychological flexibility level in bipolar disorder patients.
  Personal Information Form, Psychological Flexibility Scale pre-tests will be applied to the patients in the intervention group before the training. Afterwards, acceptance and stability-based psychoeducation consisting of 8 modules will be applied. Post-tests will be administered after the sessions, and a follow-up test will be administered one month later (at the 12th week). Psychological Flexibility Scale minimum score=28, maximum score=196. High scores indicate high psychological flexibility of individuals. The results will be evaluated in line with the data obtained.

SECONDARY OUTCOMES:
The effect of psychoeducation based on acceptance and commitment therapy on impulsivity level in bipolar disorder patients | up to 12 weeks
  The effect of psychoeducation based on acceptance and commitment therapy on impulsivity levels in bipolar disorder patients.
  Personal Information Form, Barratt Impulsivity Scale-11 Short Form pre-tests will be applied to the patients in the intervention group before the training. Afterwards, acceptance and stability-based psychoeducation consisting of 8 modules will be applied. Post-tests will be administered after the sessions, and a follow-up test will be administered one month later (at the 12th week). The Barratt Impulsivity Scale, the first and original name of the scale, has a minimum score=15 and a maximum score=60. High scores indicate high impulsivity level of individuals. The results will be evaluated in line with the data obtained.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No